CLINICAL TRIAL: NCT04989556
Title: Technology-Enhanced Palliative Care for Cancer Patients
Brief Title: Technology-Enhanced Palliative Care for Advanced Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-1052; NCI-2020-07465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1052 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-07; First posted 2021-08-04 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm
MeSH Terms: interventions — Interviews as Topic; Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (standard symptom management) (Active Comparator): Patients receive standard symptom management by palliative care team once every 4 weeks for 12 weeks. Patients and caregivers also may participate in an interview with supportive care nurse over 30-45 minutes during week 8.
  Interventions: Other: Interview; Other: Palliative Therapy; Other: Quality-of-Life Assessment
- Arm II (weekly provider-initiated remote contact) (Experimental): Patients in Phase I immunotherapy trials will receive in-person clinic visits or standard remote care encounters at least once every 4 weeks and the e-ESAS and PC provider-initiated remote contact every week. Patients and caregivers may participate in an interview with supportive care nurse over 30-45 minutes during week 8.
  Interventions: Other: Interview; Other: Palliative Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (weekly provider-initiated remote contact) (Experimental): Patients in Phase I non-immunotherapy clinical trials will receive in-person clinic visits or standard remote care encounters at least once every 4 weeks and the e-ESAS and PC provider-initiated remote contact once a week. Patients and caregivers may participate in an interview with supportive care nurse over 30-45 minutes during week 8.
  Interventions: Other: Interview; Other: Palliative Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Participate in interview
Other: Palliative Therapy — Receive standard symptom management by palliative care team
  Other Names: Comfort Care; PA-Palliative Therapy; palliation; Palliative; Palliative Care; Palliative Treatment; Symptom Management; Symptoms Management
Other: Palliative Therapy — Receive provider initiated remote contact
  Other Names: Comfort Care; PA-Palliative Therapy; palliation; Palliative; Palliative Care; Palliative Treatment; Symptom Management; Symptoms Management
  Arms: Arm II (weekly provider-initiated remote contact); Arm III (weekly provider-initiated remote contact)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire
  Arms: Arm II (weekly provider-initiated remote contact); Arm III (weekly provider-initiated remote contact)

SUMMARY:
This trial investigates technology-enhanced palliative care for patients in phase I trials with cancer that has spread to other places in the body (advanced). The goal of this study is to learn if the technology-enhanced palliative care symptom-monitoring program, when combined with in-person clinic visits and standard remote care visits (by phone or video call), helps increase quality of life and care for patients with advanced cancer participating in phase 1 immunotherapy trials.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effect size of each palliative care intervention technology-enhanced palliative care, standard palliative care [SPC]) on the symptom burden of patients prior to or while on a phase I trial.

SECONDARY OBJECTIVES:

I To estimate the effect size of each palliative care intervention (TEC, SPC) on symptom burden over a 12-week period of a phase I trial.

II. To estimate the effect size of each palliative care intervention (TEC, SPC) on clinical outcomes at 6 months post-enrollment.

III. To qualitatively assess patients' and caregivers' perceptions of receiving each TEC-based palliative care (PC) Intervention.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive standard symptom management by palliative care team once every 4 weeks for 12 weeks. Patients and caregivers also may participate in an interview with supportive care nurse over 30-45 minutes during week 8.

ARM II: Patients in Phase I immunotherapy trials will receive in-person clinic visits or standard remote care encounters at least once every 4 weeks and the e-ESAS and PC provider-initiated remote contact every week. Patients and caregivers may participate in an interview with supportive care nurse over 330-45 minutes during week 8.

ARM III: Patients in Phase I non-immunotherapy clinical trials will receive in-person clinic visits or standard remote care encounters at least once every 4 weeks and the e-ESAS and PC provider-initiated remote contact once a week. In all 3 arms, follow-up communication will occur as deemed necessary by the PC team. Patients and caregivers may participate in an interview with supportive care nurse over 30-45 minutes during week 8.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Diagnosis of advanced solid tumor
* PATIENT: Oncologic plan for a phase I trial
* PATIENT: High symptom burden (defined as a score of >= 4 on at least 1 Edmonton Symptom Assessment Scale [ESAS] symptom, AND a global distress score [GDS] of >= 20)
* PATIENT: Reliable telephone and internet access
* PATIENT: Able to communicate verbally in English and provide informed consent
* CAREGIVER: Able to communicate verbally in English and provide informed consent
* CAREGIVER: Reliable telephone and internet access

Exclusion Criteria:

* PATIENT: Low symptom burden defined as scores < 4 on all ESAS symptoms OR GDS < 20
* PATIENT: Delirium (i.e. Memorial Delirium Assessment Scale > 8)
* PATIENT: No reliable telephone or internet access
* CAREGIVER: Refusal to participate in this study
* CAREGIVER: No reliable telephone or internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-05-07 (Estimated)

PRIMARY OUTCOMES:
Change in global distress score (GDS) | Baseline to 2 weeks
  Will consist of paired t-tests for the global distress score (GDS, calculated as a sum of 9 physical and psychosocial ESAS items, scored from 0-90 in which a range over 35 indicates high distress) between baseline and 2 weeks if the Edmonton Symptom Assessment Scale (ESAS) scores are approximately normally distributed. If the data are clearly not normally distributed will conduct Wilcoxon signed rank tests.

SECONDARY OUTCOMES:
Effect size of each palliative care (PC) intervention, utilizing FAMCARE-P-13 (PRO tool assessing patient satisfaction with outpatient palliative oncology care). | At 6 months after enrollment
  We will measure incremental change in the scores of patient satisfaction using FAMCARE-P13 from the baseline values.
  We also will measure the change in the scores every 4 weeks from the baseline score at time-point T0 to the 12 study weeks: weeks 4 (T4), 8 (T8), and 12 (T12). We will additionally measure at 6 months after enrollment.
Effect size of palliative care (PC) intervention, utilizing Global Distress Score (GDS) derived from Edmonton Symptom Assessment Scale (ESAS). | At 6 months after enrollment
  We will measure incremental change in the scores for GDS using ESAS, a validated score of overall symptom intensity and burden derived from the ESAS. The GDS (range 0-90) is comprised of 9 symptoms: (1) the six physical ESAS symptoms (pain, fatigue, nausea, drowsiness, appetite, shortness of breath), (2) the two psychosocial symptoms (depression, anxiety), and (3) overall sense of wellbeing..
  We also will measure the change in the scores every 4 weeks from the baseline score at time-point T0 to the 12 study weeks: weeks 4 (T4), 8 (T8), and 12 (T12). We will additionally measure at 6 months after enrollment.
Patients' and caregivers' perceptions of receiving each technology-enhanced palliative care intervention | Up to 12 weeks on phase I trial
  We will use semi-structured interviews with patients and caregivers to assess patients and caregivers' perceptions of TEC to understand the value of PC provider-initiated contact between clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04989556/ICF_000.pdf